CLINICAL TRIAL: NCT03419676
Title: Use of Hemopatch as a Sealant at the Pancreaticojejunostomy After Pancreatoduodenectomy to Prevent Postoperative Pancreatic Fistula
Brief Title: Use of Hemopatch as a Sealant at the Pancreaticojejunostomy After Pancreatoduodenectomy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hospital Miguel Servet (Other)
Collaborators: Aragon Health Science Institute (Other Government)
Responsible Party: Principal Investigator, Mario Serradilla, MD, FACS, Professor, Attending Surgeon, Hospital Miguel Servet
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: C1834-MADIT
Record Dates: First submitted 2017-12-10; First posted 2018-02-05 (Actual); Last update posted 2022-02-11 (Actual); Status verified 2022-02

CONDITIONS: Pancreatic Fistula
Keywords: Pancreatoduodenectomy; Postoperative pancreatic fistula; Sealant; Hemopatch
MeSH Terms: conditions — Pancreatic Fistula

STUDY DESIGN:
Intervention Model Description: All patient data are anonymous. Each patient who meets the selection criteria and has signed the informed consent will be entered into a database and identified by a number (from 1 to 64). The list of patient identification numbers will be in the hands of the principal investigator. After carrying out the surgery, the patient number is entered into an online computerized randomization tool ("Randomizer for clinical trials"), https://www.meduniwien.ac.at/randomizer. It is a tool of the University of Vienna in Austria, where it is registered in a study, which allows, once the patient number is entered, the randomization of the same, obtaining one of the two methods to compare (32 patients in each study group):
  1. Basic treatment: duct-to-mucosa pancreaticojejunostomy WITHOUT Hemopatch reinforcement.
  2. The same, but reinforced WITH Hemopatch.
  Once the treatment to be performed is obtained, surgery will be carried out according to the treatment obtained in the randomization.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): No reinforcement.
- Hemopatch (Experimental): Reinforcement with Hemopatch.
  Interventions: Device: Hemopatch

INTERVENTIONS:
Device: Hemopatch — Collagen patch derived from bovine dermis, coated with NHS-PEG, applied covering the pancreaticojejunostomy after pancreatoduodenectomy once the anastomosis is completed.
  Arms: Hemopatch

SUMMARY:
The objective of this study is to determine the effect of the sealant patch Hemopatch, compared to current practice without any sealant, on the decrease of the postoperative pancreatic fistula on patients undergoing pancreatoduodenectomy for benign or malignant tumors or other benign process.

DETAILED DESCRIPTION:
Pancreaticoduodenectomy (PD) is the most common surgical procedure to treat pancreatic tumors in the head of the pancreas and periampullary region, as well as benign processes such as chronic pancreatitis. Recent advances in surgical techniques and perioperative treatments have reduced perioperative mortality below 10% in high volume centers. However, PD is associated with considerable morbidity (40-58.5%) like postoperative pancreatic fistula, delayed gastric emptying, biliary fistula, postoperative hemorrhage, and pulmonary complications.

Several surgical techniques and perioperative care have been described to prevent or reduce the incidence of pancreatic fistula after PD, including reconstruction of the digestive tract with pancreaticogastrostomy, duc-to-mucosa reconstruction or pancreaticojejunostomy by intussusception, use of somatostatin and prophylactic analogues, the use of stents in the main pancreatic duct, and use of different sealants.

Although perioperative morbidity and mortality associated with PD have improved significantly over the years, even in high-volume centers, the incidence of postoperative fistula remains at 9.9-28.5%. Therefore, the ideal pancreatic reconstruction technique that prevents fistula is not yet available.

The use of sealants has been one of the approaches taken to try to reduce the rate of fistulas. Some uncontrolled or non-randomized studies have shown that the use of fibrin glue-based adhesives in combinations with felting patches can lead to a B / C grade fistula rate of 0-10%. Only 2 randomized clinical trials have been performed with fibrin glue, with opposite results in terms of significant reduction of pancreatic fistula.

Hemopatch is a patch consisting of a soft, thin and flexible pad of collagen derived from the bovine dermis, coated with NHS-PEG (pentaerythritol polyethylene glycol ether tetra-succinimidyl glutarate). It is intended to be a surgical sealant for procedures in which control of leakage by conventional surgical techniques is ineffective or impractical, making it a plausible option to use during PD in order to decrease postoperative pancreatic fistula.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for pancreatoduodenectomy by open approach, depending on the diagnosis/nature of the tumor.
* ASA score < 4.
* Male and female patients ≥ 18 and ≤ 80 years of age.
* With the consent form signed.

Exclusion Criteria:

* Patients scheduled for pancreatoduodenectomy by open approach, depending on the diagnosis/nature of the tumor.
* ASA score < 4.
* Male and female patients ≥ 18 and ≤ 80 years of age.
* With the consent form signed.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2022-02-10 (Actual)

PRIMARY OUTCOMES:
Postoperative type B and C pancreatic fistula | Up to 3 months
  Postoperative type B and C pancreatic fistula rate defined according to the International Study Group of Pancreatic Fistula criteria, measured by amylases and/or lipases levels in the perianastomotic drainage

SECONDARY OUTCOMES:
Hospital stay | Up to 3 months
  Days of duration
Stay in intensive care unit | Up to 3 months
  Days of duration
Total postoperative fistula (including type A, B, and C) | Up to 3 months
  Percentage of patients
Reoperations including interventional radiology | Up to 3 months
  Percentage of patients
Delayed gastric emptying | Up to 3 months
  Percentage of patients
Biliary fistula | Up to 3 months
  Percentage of patients
Hemorrhage | Up to 3 months
  Percentage of patients
Deep organ space complications | Up to 3 months
  Deep organ space complications
Death, irrespective of cause | Up to 3 months
  Death
Overall complications (according to Clavien-Dindo classification) | Up to 3 months
  Percentage of patients

CONTACTS AND LOCATIONS:
Overall Officials: Mario Serradilla, Principal Investigator — Hospital Miguel Servet
Locations (1):
- Mario Serradilla Martín, Zaragoza, Spain

REFERENCES:
- [Derived] Serradilla-Martin M, Paterna-Lopez S, Palomares-Cano A, Cantalejo-Diaz M, Abadia-Forcen T, Gutierrez-Diez ML, Artigas-Marco C, Serrablo-Requejo A. Polyethylene glycol-coated haemostatic patch for prevention of clinically relevant postoperative pancreatic fistula after pancreatoduodenectomy: randomized clinical trial. BJS Open. 2023 Mar 7;7(2):zrad028. doi: 10.1093/bjsopen/zrad028. PMID 37021546

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-01-25): https://cdn.clinicaltrials.gov/large-docs/76/NCT03419676/Prot_SAP_000.pdf